CLINICAL TRIAL: NCT01852435
Title: A Multi-center, Prospective, Randomized Phase III Study of the Safety and Efficacy of R-CEOP-90/R-CEOP-70 Versus R-CHOP-50 in the Treatment of Diffuse Large B-cell Lymphoma and Follicular Lymphoma Grade 3B
Brief Title: R-CEOP-90/R-CEOP-70 Versus R-CHOP-50 in the Treatment of Diffuse Large B-cell Lymphoma and Follicular Lymphoma Grade 3B
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHL-001
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Diffuse Large B-cell Lymphoma; Follicular Lymphoma Grade 3B
Keywords: diffuse large B-cell lymphoma; follicular lymphoma grade 3B
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- R-CHOP-50 (Active Comparator): R-CHOP-50 (Rituximab 375 mg/m2 d1+Cyclophosphomide 750mg/m2 d2+Adriamycin 50mg/m2 d2+vincristine 1.4mg/m2 d2+Prednisone 60 mg/m2 d2-6) every 21 days for 6 cycles, followed by Rituximab 375 mg/m2 every 21 days for 2 cycles.
  Interventions: Drug: R-CHOP-50
- R-CEOP-70 (Experimental): R-CEOP-70 (Rituximab 375 mg/m2 d1+Cyclophosphomide 750mg/m2 d2+Adriamycin 70mg/m2 d2+vincristine 1.4mg/m2 d2+Prednisone 60 mg/m2 d2-6) every 21 days for 6 cycles, followed by Rituximab 375 mg/m2 every 21 days for 2 cycles.
  Interventions: Drug: R-CEOP-70
- R-CEOP-90 (Experimental): R-CEOP-90 (Rituximab 375 mg/m2 d1+Cyclophosphomide 750mg/m2 d2+Adriamycin 90mg/m2 d2+vincristine 1.4mg/m2 d2+Prednisone 60 mg/m2 d2-6) every 21 days for 6 cycles, followed by Rituximab 375 mg/m2 every 21 days for 2 cycles.
  Interventions: Drug: R-CEOP-90

INTERVENTIONS:
Drug: R-CEOP-70
  Arms: R-CEOP-70
Drug: R-CEOP-90
  Arms: R-CEOP-90
Drug: R-CHOP-50
  Arms: R-CHOP-50

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of R-CEOP-90/R-CEOP-70 Versus R-CHOP-50 in the Treatment of Diffuse Large B-cell lymphoma and Follicular Lymphoma Grade 3B patients.

DETAILED DESCRIPTION:
The study aims to evaluate the safety and efficacy of R-CEOP-90/R-CEOP-70 Versus R-CHOP-50 in the Treatment of Diffuse Large B-cell lymphoma and Follicular Lymphoma Grade 3B patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed de novo diffuse large B-cell lymphoma or follicular lymphoma grade 3B
2. Age>=16 y.o.,<=80 y.o.
3. ECOG < 3
4. No past history of malignancy
5. Radiologically measurable disease, CT imaging in screening showing 2 or more clearly demarcated lesions with a largest diameter > 1.5 cm, or 1 clearly demarcated lesion with a largest diameter > 2.0 cm.
6. Life expectancy>6 months
7. Informed consented

Exclusion Criteria:

1. Chemotherapy before
2. Bone marrow transplantation before
3. History of malignancy
4. Active infectious disease requiring general antibiotics, anti-fungal or anti-virus therapy
5. Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
6. Primary cutaneous, CNS, mediastinal DLBCL
7. LVEF≤50%
8. Other uncontrollable medical condition that may that may interfere the participation of the study
9. Lab at enrollment(unless caused by lymphoma)

   * Neutrophile<1.5*10^9/L
   * Platelet<80*10^9/L
   * Hemoglobulin<100g/L
   * ALT or AST >2*ULN,AKP or bilirubin >1.5*ULN
   * Creatinine>1.5*ULN
10. Not able to comply to the protocol for mental or other unknown reasons
11. Pregnant or lactation
12. Active liver or biliary disease
13. If HbsAg positive, should check HBV DNA, DNA positive patients cannot be enrolled. If HBsAg negative but HBcAb positive (whatever HBsAb status), should check HBV DNA,DNA positive patients cannot be enrolled.
14. HIV infection

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2013-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2 year

SECONDARY OUTCOMES:
overall survival | 2 year
Response rate | Every 4 cycles during treatment and then every 3 months for 2 years
  21 days as one cycle
Safety as assessed using the CTCAE | Days 1 of each course and then every 3 months for 2 years
  21 days as one cycle

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, MD, PhD, Principal Investigator
Locations (12):
- China (12):
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The first hospital of China medical university, Shenyang, Liaoning
  - Shanxi Provincial Tumor Hospital, Taiyuan, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - Shandong Provincal Hospital, Jinan
  - Shanghai Ruijin Hospital, Shanghai

REFERENCES:
- [Derived] Sun R, Zheng Z, Wang L, Cheng S, Shi Q, Qu B, Fu D, Leboeuf C, Zhao Y, Ye J, Janin A, Zhao WL. A novel prognostic model based on four circulating miRNA in diffuse large B-cell lymphoma: implications for the roles of MDSC and Th17 cells in lymphoma progression. Mol Oncol. 2021 Jan;15(1):246-261. doi: 10.1002/1878-0261.12834. Epub 2020 Nov 9. PMID 33107145
- [Derived] Xu PP, Fu D, Li JY, Hu JD, Wang X, Zhou JF, Yu H, Zhao X, Huang YH, Jiang L, Liu F, Su LP, Chen ZW, Zeng QS, Chen JP, Fang MY, Ma J, Liu T, Song YP, Yu K, Li Y, Qiu LG, Chen XQ, Gu J, Yan JS, Hou M, Huang HY, Wang L, Cheng S, Shen Y, Xiong H, Chen SJ, Zhao WL. Anthracycline dose optimisation in patients with diffuse large B-cell lymphoma: a multicentre, phase 3, randomised, controlled trial. Lancet Haematol. 2019 Jun;6(6):e328-e337. doi: 10.1016/S2352-3026(19)30051-1. PMID 31126528